CLINICAL TRIAL: NCT04131088
Title: "Follow-up of Midlines Placed Outside the Intensive Care Unit: What Happens Next, What Side Effects? A Multicenter Observational Study"
Brief Title: "Follow-up of Midlines Placed Outside the Intensive Care Unit: What Side Effects? An Observational Study"
Acronym: MidDATA
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC19_0073
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2021-09

CONDITIONS: Thrombosis
Keywords: Midline catheter; adverse event; catheter-related bloodstream infections; thrombosis
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Follow up of midlines — The follow-up data to be collected will be recorded on a monitoring logbook that will follow the patient (Appendix 4). The latter will be involved in the follow-up of his data insofar as he will be able to solicit the various professionals performing care on his midline in order to aim at the exhaustiveness of the filling of the book.

SUMMARY:
Midline catheter is a peripherally-inserted catheter, with the distal tip being placed into the axillary vein. For some indications, it's an alternative to the peripheral insert central catheters in case of limited venous access and infusions less than one month. The Midline catheter is poorly described in scientific literature; therefore, the aim of the study is to determinate the incidence of adverse events (Infections and thrombosis) and risk factors for patients with this device.

DETAILED DESCRIPTION:
The midline is a deep peripheral venous catheter whose insertion is between the lower and upper third of the arm and whose distal end does not extend beyond the axillary vein. It requires the identification of the vein by ultrasound which reserves its installation for professionals trained and authorized to use the ultrasound scanner.

Midline is currently indicated for intravenous treatments > 7 days and in patients with precarious venous capital. According to the manufacturer's instructions, it can be kept in place for up to 30 days, while the recommendations of the Centers disease of control specify that this period could be extended to 49 days.

Its use is expanding rapidly in France, thus meeting the needs of patients who do not require a central line and whose use of a standard peripheral venous catheter is not possible (low venous capital or treatment duration > 7 days). Its installation, essentially carried out by qualified anaesthetists, does not increase medical planning and is therefore an attractive alternative to the installation of a central catheter whose complications (thrombosis and infections) are known.

The only data on the complication rate, estimated at 1-2%, are from low-potency observational studies. In the absence of high-level evidence, most of the good practice recommendations published in 2019 are based on expert consensus.

This leads us to conduct a large-scale observational study to assess the complication rate and identify the associated factors. This study will provide professionals with reliable scientific data for the next review of good practice recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* No opposition to the study
* Patient requiring a midline

Exclusion Criteria:

* Patient in Intensive Care Unit or acute care unit.
* Patient with a contra indication to midline insertion: arterio-venous fistula, history of axillary lymph node clearance or radiotherapy in the infusion arm, presence of infectious skin lesions near the infusion area, presence of a prosthesis on the infusion arm or hemiplegic arm.
* Patient under legal protection measure
* Patient already enrolled
* Minor patient;
* Pregnant woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients concerned with this study requiring a midline for any indication and hospitalized in a department other than intensive care or intensive care.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
assess numbers of adverse events | through study completion, an average of 2 year
  catheter related infection yes/no vein thrombosis yes/no occlusion yes/no exposition time to a midline catheter

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France

REFERENCES:
- [Derived] Derouin Y, Le Thuaut A, Dauvergne J, Cinotti R, Cartron E. Complications and risk factors on midline catheters' follow-up about non-ICU patients: study protocol for a multicentre observational study (the midDATA study). BMJ Open. 2023 Jul 18;13(7):e067796. doi: 10.1136/bmjopen-2022-067796. PMID 37463802